CLINICAL TRIAL: NCT04462991
Title: COMPARISON OF CORNEAL MEASUREMENTS IN NORMAL AND KERATOCONUS EYES USING ANTERIOR SEGMENT OPTICAL COHERENCE TOMOGRAPHY AND PENTACAM HR TOPOGRAPHER
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Collaborators: Sara Tawfik (Unknown)
Responsible Party: Principal Investigator, Omar Said, Assistant professor of ophthalmology, Fayoum University
Other Study IDs: M 354
Record Dates: First submitted 2020-07-03; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: The Reliability of Corneal Topographic Measurements of Keratoconus Eyes
MeSH Terms: interventions — Corneal Topography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Weeks

INTERVENTIONS:
Diagnostic Test: corneal topography — In all patients, TCT will be measured first by WaveLight® Oculyzer™II Pentacam HR and second by The Optovue AS-OCT .

SUMMARY:
The purpose of current study is to provide a comprehensive comparison of the reliability of corneal topographic measurements between Optovue AS- OCT and a combined Scheimpflug imaging using Wavelight Oculyzer Pentacam HR in normal and keratoconus eyes.

ELIGIBILITY:
Inclusion Criteria:

* topography characteristic of keratoconus (skewed asymmetric bow-tie, inferior steep spot, etc.) and at least one clinical sign e.g., slit lamp findings of Munson's sign, Vogt's striae, Fleischer's ring, apical thinning, Rizutti's sign, etc.

Exclusion Criteria:

* are advanced complications of keratoconus such as corneal scars or hydrops.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: keratoconus patients
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Corneal measurments in KC CORNEAL MEASUREMENTS IN NORMAL AND KERATOCONUS EYES USING ANTERIOR SEGMENT OPTICAL COHERENCE TOMOGRAPHY AND PENTACAM HR TOPOGRAPHER | we will recruit patients who meer the inclusion criteria during the study period januray-August 2020
  In all patients, TCT will be measured first by WaveLight® Oculyzer™II Pentacam HR and second by The Optovue AS-OCT .
  KERATOCONUS EYES USING ANTERIOR SEGMENT OPTICAL COHERENCE TOMOGRAPHY AND PENTACAM HR TOPOGRAPHER

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP